CLINICAL TRIAL: NCT03382054
Title: Frailty and Post-operative Complications in Older Surgical Patients: The Implication of Frailty and Preoperative Risk Assessment - A Retrospective Analysis
Brief Title: Frailty and Post-operative Complications in Older Surgical Patients: The Implication of Frailty and Preoperative Risk Assessment
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Clinical director of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charite University, Berlin, Germany
Other Study IDs: FrailAmb II
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Frailty; Surgery; Older Patients
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Older robust surgical patients: Male and female patients with age 65 years and above scheduled for surgery, which are robust according to Fried's Modified Frailty Score.
- Older pre-frail surgical patients: Male and female patients with age 65 years and above scheduled for surgery, which are pre-frail according to Fried's Modified Frailty Score.
- Older frail surgical patients: Male and female patients with age 65 years and above scheduled for surgery, which are frail according to Fried's Modified Frailty Score.

SUMMARY:
Frailty is prevalent in older adults and may be a better predictor of post-operative morbidity and mortality than chronological age. Preoperative risk factors and physiological reserves were assessed on patients more than 70 years old who are scheduled for surgery under general or regional anesthesia. The aim of this retrospective analysis was to examine the impact of relevant geriatric assessments on adverse outcomes in older surgical patients.

DETAILED DESCRIPTION:
The goal of this study is to analyze the effect of frailty status on postoperative outcomes. These include postoperative complications (only ICD-10 coded diagnoses), length of hospitalization (ward/ICU), disposition, and survival. The project will also attempt to find synergism between a positive frailty status and common medical conditions (e.g. diabetes, congestive heart failure, coronary artery disease, dementia, and kidney disease), as well as anesthesiological and surgical processes (e.g. duration and type of anesthesia, surgical risk, and surgical discipline). Different assessment tools will be analyzed regarding their predictive power and clinical practicability. This should help improve preoperative risk assessment and allow for the multidimensional (physical, cognitive, social) identification of relevant frailty characteristics in the perioperative setting. All outcome parameters, including admission and discharge periods, will be collected using coded information from our hospital database. There will be no follow-up measurements after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age 70 years and above scheduled for surgery in the Department of Anesthesiology and Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Male and female patients with age 70 years and above scheduled for surgery
Sampling Method: Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 06/2016-12/2022
  ICD-10 coded diagnoses for the hospitalization

SECONDARY OUTCOMES:
Duration of Hospital stay | 06/2016-12/2022
Duration of Intensive Care Unit Stay | 06/2016-12/2022
Procedures | 06/2016-12/2022
  The procedures are measured regarding the following practices: anesthesiological, surgical, physiotherapeutic, social, cognitive, therapeutic, behavioral
Morbidity | 06/2016-12/2022
Ventilation | 06/2016-12/2022
  Ventilation is measured in hours.
Requirements for intensive care unit | 06/2016-12/2022
Intensive care unit scores | 06/2016-12/2022
Disease severity | 06/2016-12/2022
Postoperative Delirium | 06/2016-12/2022
  Delirium is measured with validated delirium scores.
Mortality | 06/2016-12/2022
  Mortality is measured in hospital.
Medical costs | 06/2016-12/2022
  Costs incurred during hospitalization
Physiotherapy | 06/2016-12/2022
  Physiotherapy is measured by Physiotherapists support.
Nutritional therapy 1 | 06/2016-12/2022
  Nutritional consultations
Nutritional therapy 2 | 06/2016-12/2022
  Feeding
Post - intensive care syndrome | 06/2016-12/2022
  Post - Intensive care syndrome is measured by a cluster of symptoms that are unique to the Intensive care unit environment.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No